CLINICAL TRIAL: NCT06107192
Title: Gut Microbial Metabolites Of Apple Polyphenols: Interrogating Individual Differences To Establish Functional Biomarker Utility
Brief Title: Gut Microbial Metabolites of Apple Polyphenols
Acronym: GutMMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: MaineHealth (Other); University of Hawaii Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-05787; 2022-67017-41032 (Other Grant/Funding Number: U.S. Department of Agriculture)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Controlled Feeding Trial
Keywords: Gut microbiome; Flavonoids; Isoflavones; Catechin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the crossover trial of two diets, participants will receive the same foods during both arms. The intervention and control will be delivered by a beverage containing either the active component or a nutritionally equivalent control beverage with similar flavor. Participants will not be told the order of study arms they receive. Drinks will be labeled with a code by a different researcher than the team interacting with participants. The statistician will not know which code corresponds to which intervention until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple catechin (Experimental): A 3-day controlled diet
  Interventions: Other: Dietary intervention - apple catechin diet
- Low catechin (Placebo Comparator): A 3-day controlled diet
  Interventions: Other: Dietary intervention - low catechin diet

INTERVENTIONS:
Other: Dietary intervention - apple catechin diet — The intervention will provide a catechin-containing apple juice, for consumption alongside a low catechin diet tailored to participants calorie needs for weight maintenance.
  Arms: Apple catechin
Other: Dietary intervention - low catechin diet — The intervention will provide a nutritionally-matched beverage without catechins, for consumption alongside a low catechin diet tailored to participants calorie needs for weight maintenance.
  Arms: Low catechin

SUMMARY:
The goal of this controlled feeding trial is to learn about the metabolism of polyphenols, a common class of compounds found in plant-based foods, by the gut microbiome. It will evaluate how differences in gut bacteria across individuals influence metabolism of polyphenols from foods, which may influence health benefits that people receive from different foods.

DETAILED DESCRIPTION:
This is a randomized, cross-over controlled feeding trial. Thirty healthy adult volunteers will be selected to participate on the basis of urinary screening results measuring a gut bacterial metabolite that is produced following consumption of a soy food: 15 O-desmethylangolensin (ODMA) producers and 15 age and gender-matched ODMA non-producers will be included. Participants will be assigned to consume two diets in random order: an apple catechin diet that provides a controlled amount of catechins in apple juice, and a nutritionally-matched low catechin diet. Both diet phases will last 3 days, with a 10 day washout period in between the two diet phases.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Any gender identification, aged 18 - 45.
4. BMI 18.5 - 40 kg/m^2
5. Ability to consume the intervention foods and beverages and be willing to adhere to the dietary regimen.
6. Agreement to provide urine and fecal samples according to the study protocol.
7. Agreement to adhere to avoid high catechin foods (tea, chocolate) for 4 weeks.
8. Able to come to the study location for 8 visits according to the study schedule.
9. As assessed through an initial urine screening phase, a person is eligible either on the basis of (1) the presence of a urinary marker for soy isoflavone metabolism (ODMA), or (2) as a control matched for age and gender.

Exclusion Criteria:

1. Current, regular use of antacids or acid reducers.
2. Systemic antibiotic use within the past month prior to the urinary screening until completion of the dietary intervention.
3. Pregnancy or lactation, within 3 months post-partum (regardless of breastfeeding) at screening or planning to become pregnant during the study duration.
4. Known allergic reactions to components of the foods or beverages of the study diet (soy, wheat, dairy, peanut, tree nuts, apples, eggs) or any history of anaphylactic food allergy.
5. Current diagnosis of renal, hepatic, or gastrointestinal conditions.
6. History of stroke.
7. Underweight (BMI <18.5 kg/m^2) or severe obesity (BMI >40 kg/m^2).
8. Under 18 years or above 45 years of age.
9. Unwilling or unable to participate in the controlled dietary intervention or provide urine or fecal samples.
10. Has a pacemaker, implanted defibrillator, or other implanted electronic device.
11. Change of body weight >10% between screening and dietary intervention.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Mean sum catechin metabolites | Post 3-day intervention vs. post 3-day control
  Mean difference in sum catechin metabolite concentration in response to the intervention, stratified by ODMA producers and non-producers.

SECONDARY OUTCOMES:
Mean individual catechin metabolites | Post 3-day intervention vs. post 3-day control
  Mean differences in individual valerolactone and valeric acid concentrations in response to the intervention, stratified by ODMA producers and non-producers.
Differences in microbiome profiles | Post 3-day intervention vs. post 3-day control
  Differences in microbiome profiles in response to the 3-day intervention.
Difference in microbiome diversity | Post 3-day intervention vs. post 3-day control
  Differences in microbiome diversity in response to the 3-day intervention.
Difference in microbial species abundance | Post 3-day intervention vs. post 3-day control
  Differences in microbial species abundance in response to the 3-day intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Slavin, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Department of Nutrition and Food Science, College Park, Maryland, United States